CLINICAL TRIAL: NCT04285073
Title: Prospective, Multicenter, Non-randomized, Single Arm Clinical Trial to Evaluate the Safety and Efficacy of e-PTFE Grafts Inner Surface-treated With Paclitaxel as an Access for Hemodialysis in Patients With End-stage Renal Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Kim Dae Joong, professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SMC 2018-03-017
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Hemodialysis Access Failure
Keywords: hemodialysis; vascular access; arteriovenous graft; paclitaxel-eluting graft

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paclitaxel-eluting graft (Experimental): Single-arm
  Interventions: Device: Paclitaxel-eluting graft

INTERVENTIONS:
Device: Paclitaxel-eluting graft — Implantation of e-PTFE Grafts inner surface-treated with paclitaxel as access for hemodialysis

SUMMARY:
This prospective, multicenter, non-randomized, single-arm Clinical trial aims to evaluate the safety and effectiveness of the use of paclitaxel-coated arteriovenous graft (AVG) on the inner wall of ePTFE graft, which is designed to reduce neointimal hyperplasia that causes stenosis and thrombosis after implantation of AVG.

DETAILED DESCRIPTION:
1. Evaluation of safety Primary outcome: all adverse events occurring in the subject
2. Evaluation of effectiveness Primary outcome: AV graft primary patency Secondary outcome: AV graft secondary patency

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female between the ages of 20 and 80
* Patients currently undergoing or scheduled for hemodialysis due to end-stage kidney disease.
* Patients who decided to receive AVG procedure in forearm due to inability to perform autologous arteriovenous fistula (AVF)
* Patients with a high risk of stenosis (neointimal hyperplasia) or thrombosis when artificial blood vessels were implanted

Exclusion Criteria:

* Pregnant or lactating women
* Patients who are currently diagnosed with malignant tumors and are receiving chemotherapy or radiotherapy
* Patients with life expectancy less than 12 months
* Patients expected to receive a kidney transplant during the trial
* Patients with current or suspected infection
* Acute psychiatric problems require treatment
* Patients who have inserted a catheter into an artery or vein in their upper limb for AVG procedure within the last 30 days
* Patients with coagulation disorder, platelet count <50,000 / Ul
* Patients with a neutrophil count of less than 1,500 cells / mm3
* Patients judged to be unable to insert grafts by the operator

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-11-13 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Up to 2 years after implantation of AVG
  All adverse events occurring in the subject
Primary patency | at 6 months after implantation of AVG
  Percentage of no intervention (intravascular or surgical) to maintain or recover blood flow or occurrence to access thrombosis

SECONDARY OUTCOMES:
Secondary patency | Up to 2 years after implantation of AVG
  Percentage of no permanent failure of AVG

CONTACTS AND LOCATIONS:
Overall Officials: Dae Joong Kim, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea